CLINICAL TRIAL: NCT03275857
Title: A Pilot Study of Cisplatin in Castration Resistant Prostate Cancer That is Becoming Refractory to Enzalutamide
Brief Title: Cisplatin in Castration Resistant Prostate Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Roswell Park Cancer Institute (Other)
Responsible Party: Principal Investigator, Deepak Sahasrabudhe, Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UGUP-17050
Record Dates: First submitted 2017-07-27; First posted 2017-09-08 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cisplatin (Other)
  Interventions: Drug: Cisplatin

INTERVENTIONS:
Drug: Cisplatin — Weekly IV

SUMMARY:
It is hypothesized that treatment with cisplatin will reverse emerging refractoriness to enzalutimide in patients with CRPC by affecting AR function.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of prostate cancer
* Age 18 yrs or older
* Able to provide written, informed consent
* Subjects who have received docetaxel for metastatic disease are eligible if absolute neutrophil count is greater than 100 and platelet count is greater than 100,000 and their bone marrow reserve is deemed to be adequate
* Subjects with castration resistant prostate cancer, as defined by having testosterone level of less than 50 Nano gram/dl, being treated with enzalutamide with a rise in PSA, confirmed with a repeat measurement within 1 to four weeks, or asymptomatic radiographic progression

Exclusion Criteria:

* Subjects with estimated glomerular filtration rate of less than 50 ml/min
* Subjects with hearing impairment. The treating physician may decide which subjects should not receive cisplatin based on audiometry or based on clinical judgment.
* Subjects with grade 2 or greater neuropathy
* Subjects who in the opinion of the treating physician could not tolerate the standard hydration before receiving cisplatin
* Chemotherapy naïve subjects who in the opinion of the treating physician should receive docetaxel instead of enrolling on the trial and receive cisplatin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-09-21 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Response to dosing differences of Cisplatin from lab and scan results | 2 years
  Measures of response will be decline in Prostate Specific Antigen (PSA) and regression of metastases.
Toxicity observed with dosing differences of Cisplatin | 2 years
  Blood samples and physical assessments will be conducted and reviewed to determine toxicity of treatment. Toxicity would be symptoms such as ringing in the ears (tinnitus) peripheral neuropathy or lab findings such as rise in creatinine, electrolyte abnormalities such as low magnesium.

CONTACTS AND LOCATIONS:
Locations (1):
- Wilmot Cancer Institute, Rochester, New York, United States